CLINICAL TRIAL: NCT03243162
Title: Improving ACL Reconstruction Outcomes: Cognitive-Behavioral Based Physical Therapy
Brief Title: Improving ACL Reconstruction Outcomes: CBPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kristin Archer, Associate Professor and Vice Chair of Research, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 161927
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: ACL Injury; ACL - Anterior Cruciate Ligament Rupture; ACL Sprain; ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBPT-ACLR (Experimental): CBPT-ACLR program consisting of weekly phone calls.
  Interventions: Behavioral: CBPT-ACLR
- Education (Active Comparator): Education program consisting of weekly phone calls.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: CBPT-ACLR — The CBPT-ACLR program focuses on improving sports function and return to sport. CBPT-ACLR sessions cover realistic expectations, relaxation strategies, problem-solving training, cognitive restructuring, and behavioral self-management (i.e., graded activity, goal setting, managing setbacks and symptom management plans). Each session builds upon the content of the previous session using an action plan and weekly homework is personally tailored based on patient goals. The program consists of one preoperative telephone session and six postoperative telephone sessions with a physical therapist. Each patient randomized into the CBPT-ACLR program will receive a manual to follow along with the study therapist.
  Arms: CBPT-ACLR
Other: Education — The education program focuses on postoperative ACLR recovery. Sessions address benefits of physical therapy, proper biomechanics during sports and other functional activity, importance of early exercise after surgery, and ways to promote healing. Education on stress reduction, sleep hygiene, energy management, communication with health providers, and preventing future injury are also provided. The Education program is matched to the CBPT-ACLR treatment in terms of session frequency, length and contact with the study therapist. Each patient randomized into the Education program will receive a manual to follow along with the study therapist.
  Arms: Education

SUMMARY:
The overall objective of this study is to conduct a two-group randomized trial to examine the efficacy of cognitive-behavioral based physical therapy (CBPT) for improving knee function, return to sport, and quality of life outcomes in patients following ACL reconstruction (ACLR). The study consists of two treatment groups: telephone-based cognitive-behavioral based physical therapy for ACLR (CBPT-ACLR) and telephone-based Education. The central hypothesis is that the CBPT-ACLR participants relative to the Education group will demonstrate significantly greater improvement in postoperative outcomes at 12 months following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking (due to feasibility of employing study personnel to deliver and assess the study intervention);
2. 14 to 35 years of age (children 14 and older have skeletal maturity and adults 35 and younger are less likely to have symptoms of knee osteoarthritis);
3. no previous surgery to either knee;
4. time from injury to surgery 12 months or less;
5. active participation in a sport on a weekly basis prior to injury

Exclusion Criteria:

1. bilateral simultaneous ACL reconstructions;
2. revision ACLR;
3. any concurrent ligament (MCL, LCL, or PCL) surgical procedures;
4. concurrent osteotomies or meniscus transplantations;
5. surgery secondary to trauma, tumor, or infection;
6. having workman's compensation insurance for surgery;
7. on active military duty;
8. medical history of schizophrenia or other psychotic disorder; and
9. unable to provide stable address and access to a telephone

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) sport and recreation sub-scale | Up to 12 months after ACLR surgery
  knee function relating to sport/recreation
Marx Activity Rating Scale | Up to 12 months after ACLR surgery
  The Marx Activity Rating Scale measures knee function relating to running, cutting, decelerating, and pivoting.

SECONDARY OUTCOMES:
Subjective Patient Outcome for Return to Sports (SPORTS) | Up to 12 months after ACLR surgery
  The SPORTS score measures 1) ability to perform the same sport with the same level of effort, 2) ability to reach the same level of performance, and 3) ability to perform with no pain or in spite of the pain.
Knee Injury and Osteoarthritis Outcome Score (KOOS) knee related quality of life sub-scale | Up to 12 months after ACLR surgery
  knee function relating to quality of life
EQ-5D | Up to 12 months after ACLR surgery
  The EQ-5D is used to measure non-disease-specific quality of life and calculate cost-effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Archer, PhD, DPT, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Cleveland Clinic, Garfield Heights, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee